CLINICAL TRIAL: NCT06923501
Title: Feasibility, Acceptability, and Preliminary Outcomes of a Mobile App for Coping With Cancer
Brief Title: Evaluation of a Mobile App Program for Coping With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000037763
Record Dates: First submitted 2025-03-23; First posted 2025-04-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: mobile application; app; cancer; coping; quality of life; distress
MeSH Terms: conditions — Neoplasms; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile App Intervention (Experimental): Participants will be asked to use the 13-session Coping with Cancer Program in a mobile app.
  Interventions: Device: Tools for Coping with Cancer Calm Health mobile app program

INTERVENTIONS:
Device: Tools for Coping with Cancer Calm Health mobile app program — Participants will be asked to use a 13-session self-management program "Tools for Coping with Cancer" within the Calm Health mobile app.

SUMMARY:
The goal of this clinical trial is to learn if a mobile app program for people with a history of cancer can help treat distress. The main questions it aims to answer is:

Do participants use the Tools for Coping with Cancer Calm Health mobile app and do they find it helpful?

Does the Tools for Coping with Cancer Calm Health mobile app improve mood, quality of life, and help with coping?

Participants will be asked to use a 13-session self-management program (Tools for Coping with Cancer) housed within the Calm Health app. Participants will use this app on their own device, in their own home. Participants will have access to the program for 8 weeks and will be asked to work their way through the program at their own pace. Participants will be asked to complete questionnaires about their mood, quality of life, coping, and experience with the app three times: at the start of the study, after 8 weeks using the app, and then 3-months after using the app.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility, acceptability, and preliminary effectiveness of a self-management mobile app on mood, quality of life, psychological flexibility, and adaptive coping in a population of people with cancer.

The intention of this research is to meet the most common unmet supportive care needs such as anxiety and depression, pain, insomnia, and fear of cancer recurrence utilizing evidence-based intervention that is accessible and self-paced.

We hypothesize that the Tools for Coping with Cancer mobile app program will:

1. Be feasible and acceptable to participants, as rated by interest, accrual, and completion rates, acceptability ratings, and participant satisfaction with the program.
2. Have a statistically significant effect on symptoms of depression, anxiety, psychological flexibility, adaptive coping, and quality of life. We further hypothesize that these improvements will be retained at 3-months post-intervention.

The primary objective is to determine the feasibility and acceptability of a self-management mobile app intervention as measured by participant interest, accrual, completion, satisfaction, acceptability, and app usage.

The secondary objective is to evaluate preliminary outcomes related to mood, quality of life, psychological flexibility, and adaptive coping, and will be measured using self-report questionnaires.

This is a prospective pilot feasibility, acceptability, and effectiveness study.

The intervention is a 13-session self-management program housed within the Calm Health app. Participants will have access to the program for 8 weeks and will be asked to work their way through the program at their own pace.

Participants will complete a series of self-report surveys to evaluate the primary and secondary objectives of the study. Additionally, researchers will have access to data reporting participant's usage patterns of the app, including the frequency and duration of session play.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study (8 weeks active intervention and 3-month follow up)
* Have a confirmed diagnosis of cancer; or have been treated for cancer within the last two years, including adjuvant therapies
* Over the age of 18
* Able to understand and read English
* Able to navigate a mobile app with minimal assistance from study staff
* Able to provide informed consent

Exclusion Criteria:

* Are taking part in psychotherapy at any time during the study
* Have an un-treated or under-treated mental health disorder based on pre-study screening that may require a referral to individual mental health care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Participant interest | Up to 12 months
  The number of individuals who initiate evaluating eligibility.
Accrual | Up to 12 months
  The number of individuals who provide consent.
Participant completion | Up to 12 months
  The number of individuals who complete all sessions of the program.
Participant satisfaction | Up to 18 months
  A Likert-type scale ranging from very dissatisfied to very satisfied on the program overall as well as each session.
  Minimum value: 0 (not at all satisfied) Maximum value: 140 (Very satisfied with the program as a whole; very satisfied with each individual session) Lower numbers indicate worse outcome.
Helpfulness | Up to 18 months
  A Likert-type scale ranging from very unhelpful to very unhelpful on the program overall as well as each session.
  Minimum value: 0 (not at all helpful) Maximum value: 140 (Found program as a whole and each individual session very helpful).
  Lower numbers indicate worse outcome.
Acceptability | Up to 18 months
  A 10-item acceptability questionnaire (Theoretical Framework of Acceptability) evaluating affective attitude, burden, ethicality, perceived effectiveness, intervention coherence, self-efficacy, opportunity costs, and general acceptability.
  Minimum value: 0 Maximum value: 100 Higher score indicates greater acceptability
Usage | Up to 18 months
  Participant usage of the app, including frequency and duration of session play will be captured.

SECONDARY OUTCOMES:
Depression | Up to 18 months
  Will be measured using:
  Patient Health Questionnaire-9; a 9-item scale evaluating the frequency of depression symptoms over a two week period.
  Minimum score: 0 Maximum score: 27 Higher score = worse outcome
Anxiety | Up to 18 months
  Will be measured using:
  Generalized Anxiety Disorder-7; a 7-item scale evaluating the frequency of anxiety symptoms over a two week period.
  Minimum score: 0 Maximum score: 21 Higher score = worse outcome
Adaptive Coping | Up to 18 months
  Will be measured using the Brief COPE, a 28-item measure of coping in response to stressful situations.
  Minimum score: 28 Maximum score: 112 Outcome depends on the score of each subscale, of which there are 14. Some subscales reflect adaptive coping, while others reflective maladaptive coping.
Health Related Quality of Life | Up to 18 months
  Will be measured by the FACT-G (Functional Assessment of Cancer Therapy, General), a 27-item questionnaire designed to measure four domains of health related quality of life in people with cancer: Physical, social, emotional, and functional well-being.
  Minimum score: 108 Maximum score: 0 Higher scores indicate better outcome
Psychological Flexibility | Up to 18 months
  Will be measured by the Brief Experiential Avoidance Questionnaire, a 15-item questionnaire measuring willingness to remain in contact with distressing emotions, memories, thoughts, and physical sensations.
  Minimum score: 15 Maximum score: 90 Higher scores indicate worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Cartagena, PhD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No
Study limited to one site. No need to share data.

REFERENCES:
- [Background] Agboola SO, Ju W, Elfiky A, Kvedar JC, Jethwani K. The effect of technology-based interventions on pain, depression, and quality of life in patients with cancer: a systematic review of randomized controlled trials. J Med Internet Res. 2015 Mar 13;17(3):e65. doi: 10.2196/jmir.4009. PMID 25793945